CLINICAL TRIAL: NCT07232277
Title: Intraoperative Venous Congestion and Cardiac Surgery-associated Acute Kidney Injury (CSA-AKI): a Prospective Cohort Study
Brief Title: Venous Congestion and Cardiac Surgery-Associated Acute Kidney Injury
Status: Recruiting | Type: Observational
Sponsor: Zhuan Zhang (Other)
Responsible Party: Sponsor-Investigator, Zhuan Zhang, MD, the Deputy Director of Anesthesiology, the Affiliated Hospital of Yangzhou University, Yangzhou University, Yangzhou University
Organization: Yangzhou University (Other)
Other Study IDs: 20240916
Record Dates: First submitted 2024-12-02; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Intraoperative; Venous Congestion; Cardiac Surgery-associated Acute Kidney Injury
MeSH Terms: conditions — Hyperemia | interventions — Comorbidity; Laboratories

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant: Adult patients scheduled to undergo elective cardiac surgery
  Interventions: Other: collection of demographic characteristics and comorbidities; Other: surgery-related parameters and kidney function assessments; Other: collection of biological (laboratory) parameters; Other: collection of hemodynamic parameters; Other: collection of echocardiographic parameters and venous ultrasound assessments

INTERVENTIONS:
Other: collection of demographic characteristics and comorbidities — 1. gender, age, BMI, ASA classification, NYHA (New York Heart Association) classification.
  2. smoking history, medical history (hypertension, diabetes mellitus, Hyperlipidemia, stroke, anaemia, chronic obstructive pulmonary disease, pulmonary hypertension, preoperative atrial fibrillation, peripheral artery disease), preoperative ACEI, ARB, beta-blockers, loop diuretics, contrast agent, aspirin, and spironolactone use.
Other: surgery-related parameters and kidney function assessments — 1. surgery type, surgery duration, CPB duration, aortic cross-clamp duration, blood loss, intraoperative fluid infusion, intraoperative urine output, intraoperative blood transfusion, intraoperative anesthetics and vasoactive medications.
  2. baseline and postoperative eGFR, duration of mechanical ventilation, duration of vasopressor support, postoperative CRRT initiation, major bleeding, deep sternal wound infection/mediastinitis, surgical re-intervention, ICU LOS, hospital LOS, postoperative stroke, postoperative delirium, complications up to 30 days after surgery, 30-day inpatient mortality, survival status at discharge, and one year follow-up.
  3. a composite endpoint of major complications after surgery defined as at least one of the following: death, prolonged ventilation (>24 h), stroke, severe AKI, deep sternal wound infection, and reoperation for any reason.
  4. CSA-AKI diagnosed using the KDIGO criteria.
  5. acute kidney disease assessment.
  6. major adverse kidney events.
Other: collection of biological (laboratory) parameters — 1. WBC, CRP, IL-6, IL-1β, TNF-α, serum Amyloid A, procalcitonin, catecholamines, cortisol, SOD.
  2. creatinine, uric acid, BUN, CysC, β2-MG, eGFR.
  3. CK-MB, high-sensitivity troponin, NT pro-BNP, BNP.
  4. hemoglobin, hematocrit, sodium, arterial lactate, liver enzymes.
Other: collection of hemodynamic parameters — 1. blood pressure, heart rate, CVP;
  2. CO, CI, SV, SVI,SVV;
  3. intra-abdominal pressure;
  4. vasoactive drug doses in the first hour in the ICU.
Other: collection of echocardiographic parameters and venous ultrasound assessments — 1. Left ventricle systolic function, including LVOT, LVEF, MPI; left ventricular diastolic function, including mitral flow-derived Doppler indices, pulmonary vein Doppler indices.
  2. Right ventricular systolic function, including TAPSE. Right ventricular diastolic function, inferred from an hepatic vein flow in the absence of a dysrhythmia or pacing.
  3. Inferior vena cava (IVC) measurements.
  4. Hepatic vein Doppler parameters.
  5. Portal vein Doppler parameters.
  6. Renal vein Doppler parameters.
  7. Renal artery blood flow Doppler parameters.

SUMMARY:
Venous pressure is often overlooked as an important hemodynamic parameter. Elevated venous pressure and blood stasis in organ tissues can lead to interstitial edema. Intraoperative venous blood stasis can rapidly increase interstitial pressures within organ tissues, especially in organs encapsulated by tissue envelopes, such as the kidney, thereby rapidly reducing effective circulating blood flow to the organ. Systemic venous blood stasis, which tends to occur in patients with right heart failure or pulmonary hypertension, as well as in patients with fluid overload, can lead to intraoperative stasis in multiple organs and tissues, mediating the development of multisystem complications, including acute kidney injury. Therefore, timely, effective, and accurate intraoperative assessment of systemic venous blood stasis is particularly important.

When right heart failure and/or volume overload occurs in the body, changes in right atrial pressure are transmitted to the venous system of organs throughout the body, with dilatation of the inferior vena cava (IVC), obstruction of blood return from the hepatic, portal, and renal veins, and abnormal venous flow signals and altered ultrasound Doppler flow patterns.

The primary objective of this prospective cohort study is to explore if intraoperative systemic venous congestion during cardiac surgery is associated with postoperative CSA-AKI. In doing so, we seek to identify a promising physiological marker that can provide cues for the prediction of CSA-AKI. This study will also investigate the relationship between intraoperative systemic venous congestion and postoperative complications, and explore the relationship between each separate venous congestion and AKI after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled to undergo elective cardiac surgery;
2. ≥ 18 years.

Exclusion Criteria:

1. Contraindications for TEE;
2. Emergency cardiac surgery;
3. Major vascular surgery;
4. Redo cardiac surgery;
5. Abnormal preoperative renal function;
6. Severe chronic kidney disease (estimated glomerular filtration rate < 15 ml/min/1.73 m2 or dialysis);
7. History of kidney transplantation;
8. Severe infection requiring continuous antibiotic therapy；
9. Severe preoperative heart failure with left ventricular ejection fraction < 30%;
10. A critical preoperative state (mechanical circulatory support, extracorporeal membrane oxygenation, current renal replacement therapy [RRT], mechanical ventilation, or cardiac arrest necessitating resuscitation);
11. Multi-organ dysfunction;
12. Known conditions that may interfere with the assessment or interpretation of hepatic vein, portal vein blood flow (such as liver cirrhosis or portal vein thrombosis) or the renal vein blood flow and renal artery blood flow (such as urinary tract obstruction);
13. Planned cardiac transplantation or ventricular assist device implantation;
14. Pregnancy;
15. Insufficient ultrasonographic imaging;
16. Restarting CPB after first CPB cessation during surgery;
17. Requirement for cardiac assist devices (ECMO, IABP, or ventricular assist device) after CPB intraoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo elective cardiac surgery
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury defined by an increase in serum creatinine of ≥150% of baseline or an elevation of 0.3 mg/dL or more within a contiguous period of 48 hours. (KDIGO criteria) | 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Zhang, MD, Principal Investigator — The Department of Anesthesiology, The Affiliated Hospital of Yangzhou University, Yangzhou University
Locations (1):
- No. 368 Hanjiang Middle Road, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No